CLINICAL TRIAL: NCT07373717
Title: Consistency of Fluid Tolerance Evaluation Methods and Their Correlation With Clinical Outcomes in Shock Patients:A Prospective, Observational Study
Brief Title: Consistency of Fluid Tolerance Evaluation Methods and Their Correlation With Clinical Outcomes in Patients With Shock
Status: Enrolling by invitation | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Professor, Southeast University, China
Other Study IDs: 20251107 fluid management
Record Dates: First submitted 2025-12-29; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Shock
Keywords: VExUS; Fluid Resuscitation; Fluid Responsiveness; Fluid Overload; Shock
MeSH Terms: conditions — Shock; Edema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to explore the feasibility and scientific validity of carotid-jugular Doppler in evaluating volume tolerance in shock patients (with the VExUS score as an important reference standard), and to conduct an in-depth analysis of the correlation between its monitoring indicators and patient prognosis.The primary endpoint is comparison of the agreement between hands-free carotid-jugular Doppler and the VExUS score in evaluating volume tolerance.The secondary endpoint is correlation between volume tolerance assessed by hands-free carotid-jugular Doppler and the clinical outcomes of shock patients.

ELIGIBILITY:
Inclusion Criteria:

* Shock patients admitted to the ICU are defined as those with persistent hypotension (systolic blood pressure < 90 mmHg or a decrease of ≥ 40 mmHg from the baseline blood pressure) accompanied by signs of tissue hypoperfusion.
* Age ≥ 18 years old.
* The patient or their legal representatives signed the informed consent form.

Exclusion Criteria:

* Patients with severe pulmonary circulatory disorders such as severe pulmonary hypertension and acute pulmonary embolism.
* Patients with right ventricular myocardial infarction or severe tricuspid regurgitation.
* Patients with severe neck trauma or deformity that affects Doppler examination of cervical arteries and veins, or those with anatomical contraindications preventing evaluation of at least one cervical artery or vein.
* Pregnant or lactating women.
* Patients with diseases that may interfere with abdominal ultrasound examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-11-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Hands-free Carotid Artery and Vein Doppler Parameters | Time of shock in ICU within 3 days
  Elevate the patient's upper body to 45°, keep the legs flat, place the long axis of the probe perpendicular to the carotid vessels (with the probe height not exceeding the upper edge of the thyroid cartilage), locate the optimal signals of the common carotid artery and internal jugular vein waveforms, and then fix the probe.

SECONDARY OUTCOMES:
PiCCO | Time of shock in ICU within 3 days
  Inject cold saline through central venous catheterization, sense temperature changes via arterial catheter, and obtain hemodynamic parameters such as cardiac output by combining thermodilution and pulse contour analysis.
Venous Excess Ultrasound Score | Time of shock in ICU within 3 days
  Evaluate the diameter, waveform, etc. of the inferior vena cava, hepatic veins, portal vein, and intrarenal veins sequentially via ultrasound, and comprehensively derive a grade ranging from 0 to 3.Grade 0: No congestion; Grade 1: Mild congestion; Grade 2: Moderate congestion; Grade 3: Severe congestion.
Bioelectrical Impedance Analysis | Time of shock in ICU within 3 days
  Attach electrodes to the patient's limbs, input basic information, measure impedance of multiple parts with multi-frequency technology, and quickly obtain parameters such as body composition.
Duration of shock | Time of shock in ICU within 28 days
  Time of shock in ICU within 28 days
Duration of Mechanical Ventilation | up to 24 weeks
  Duration of Mechanical Ventilation During ICU Admission
Total Length of Hospital Stay | up to 24 weeks
  Total Length of Hospital Stay
Length of ICU stay | up to 24 weeks
  Length of ICU stay
mortality of 28 days | Incidence of death during 28 days
  Incidence of death during 28 days
In-hospital Mortality | up to 24 weeks
  In-hospital Mortality
Vasoactive Agent Dosage | up to 24 weeks
  Vasoactive Agent Dosage During ICU Admission
Time without vasoactive agents within 28 days | Time without vasoactive agents within 28 days
  Time without vasoactive agents within 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital Affiliated to Southeast University, Nanjing, Jiangsu, China